CLINICAL TRIAL: NCT04733170
Title: Clinical Performance Evaluation of KnowNow SARS-CoV-2 Test for the Detection of COVID-19 Antigen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vatic Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: VATIC-0101
Record Dates: First submitted 2021-01-22; First posted 2021-02-01 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: KnowNow SARS-CoV-2 Rapid Antigen Test — KnowNow SARS-CoV-2 Rapid Antigen Test for the detection of Covid-19 in saliva, as compared to high sensitivity reverse transcription polymerase chain reaction (RT-PCR) of nasopharyngeal swabs as the reference test method

SUMMARY:
This is an international, multicentre, non-interventional, observational study to assess the clinical diagnostic performance of a rapid, point of care (POC) COVID-19 (SARS-CoV-2) antigen In vitro diagnostic (IVD), The KnowNow SARS-CoV-2 Rapid Antigen Test, using saliva samples when compared to reverse transcription polymerase chain reaction (RT-PCR) as the standard detection of COVID-19 infection.

DETAILED DESCRIPTION:
The KnowNow SARS-CoV-2 Rapid Antigen Test which uses saliva and is a lateral flow diagnostic device that can detect the SARS-CoV-2 specific Antigens that are present on the surface of the virus. The KnowNow test is an affordable, user friendly, and point of care device that can be mass produced as part of a multipronged strategy to address the global COVID-19 pandemic.

A saliva sample is collected from someone with suspected COVID-19 and mixed with a running buffer. The mixture is added to the sample pad of the KnowNow test, from where it migrates through the lateral flow strip. If COVID-19 Antigens are present, they bind to capture proteins on a test line and are made visible by secondary reagents within the device. The test result is visually assessed after 15-30 minutes and provides a binary positive (two lines) or negative (one line) result. Levels of COVID-19 Antigen differ dependent on disease progression. A visible test line (marked T) indicates the presence of COVID-19 Antigen in sufficient quantity in the collected sample to be detected. The appearance of the control line (marked C) confirms that the test has been performed correctly.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or over (or age of adult consent in some states within the United States).
2. Suspected COVID-19 infection and / or presenting with at least 1 recognised symptom Fever or chills. ie: Cough. Shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat
3. Be willing and able to comply with study procedures.
4. Be able to give written informed consent.

Exclusion Criteria:

1. Inability to give written informed consent.
2. Vaccinated against SARS-CoV-2
3. Adults unable to undertake the requirements of the nasopharyngeal or saliva sample collection for physical or psychological reasons
4. Subjects with other significant disease, condition, or at the Clinician's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female aged 18 years or over (or age of adult consent in some states within the United States) with suspected COVID -19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Assess clinical diagnostic performance of the KnowNow SARS-CoV-2 Rapid Antigen Test | 6 months
  This includes determination of the sensitivity/positive percent agreement (PPA), specificity/negative percent agreement (NPA), positive predicted value (PPV) and negative predictive value (NPV).

SECONDARY OUTCOMES:
Efficacy to assess the test compared to the reference test method | 6 months
  * Calculated Sensitivity/PPA, Specificity/NPA, PPV and NPV of the KnowNow SARS-CoV-2 Rapid Antigen Test compared to RT-PCR as SOT in individuals with and without COVID-19 symptoms.
  * Calculated Sensitivity/PPA, Specificity/NPA, PPV and NPV of the KnowNow SARS-CoV-2 Rapid Antigen Test compared to RT-PCR as the reference method in individuals with and without COVID-19 symptoms.
  * Calculated Sensitivity/PPA between the KnowNow SARS-CoV-2 Rapid Antigen Test and RT-PCR tests stratified using cycle threshold (CT) values.
Usability Questionnaire to evaluate the use of the test with 2 saliva collection methods | 6 months
  Evaluation of the 2 saliva collection methods by a patient questionnaire with responses recorded by a healthcare provider. responses are on a numerical scale graded 1 to 9. 1 = 'hard' to 9 which is 'easy'.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Sheppard, BA, Study Director — Vatic Ltd.

IPD SHARING:
Plan to Share IPD: No